CLINICAL TRIAL: NCT00683501
Title: A Phase II Study to Investigate the Safety, Efficacy, and Pharmacokinetic Profile of Twice-Daily DNB-001 in Previously Untreated Patients With Elevated Intraocular Hypertension
Brief Title: Safety, Efficacy, and Pharmacokinetic Profile of DNB-001 in Subjects With Elevated Intraocular Pressure
Acronym: DNB-001
Status: Completed | Phase: Phase 1 / Phase 2 | Type: Interventional
Sponsor: Danube Pharmaceuticals, Inc. (Industry)
Responsible Party: Mr. Clive Migdal, Western Eye Hospital
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: DNB-001-CT001; EudoraCT 2006-003907-38
Record Dates: First submitted 2008-05-21; First posted 2008-05-23 (Estimated); Last update posted 2009-06-03 (Estimated); Status verified 2009-06

CONDITIONS: Ocular Hypertension; Elevated IOP; Glaucoma
Keywords: ocular hypertension; elevated IOP; glaucoma; neuroprotection
MeSH Terms: conditions — Ocular Hypertension; Glaucoma

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes

ARMS (5):
- 1 (Experimental): dosage X mg BID
  Interventions: Drug: DNB-001
- 2 (Experimental): dosage Y mg BID
  Interventions: Drug: DNB-001
- 3 (Experimental): dosage Z mg BID
  Interventions: Drug: DNB-001
- 4 (Experimental): dosage 2Z mg BID
  Interventions: Drug: DNB-001
- 5 (Placebo Comparator): Placebo BID
  Interventions: Drug: DNB-001

INTERVENTIONS:
Drug: DNB-001 — four dosages of DNB-001, one placebo dosage

SUMMARY:
A Multi-Centre, Double-Blind, Randomised, Parallel-Group, Placebo-Controlled Phase 1I Study to Investigate the Safety, Efficacy, and Pharmacokinetic Profile of Twice-Daily DNB-001 in Previously Untreated Patients with intraocular Hypertension

DETAILED DESCRIPTION:
To evaluate the efficacy of four dosages of mg DNB-001 administered twice daily (bid) per os (p.o.) as an anti-ocular hypertensive agent, compared with placebo administered bid po, for 28 days, in patients with ocular hypertension.

ELIGIBILITY:
Inclusion Criteria:

* Male or female, at least 18 years old, in general good health, not presently treated for elevated intraocular pressure (IOP), with best corrected Early Treatment Diabetic Retinopathy Study (ETDRS) visual acuity score equivalent to a Snellen score of 20/50 or better in each eye and lOP of 21 to 29 mm Hg at baseline.

Exclusion Criteria:

* Use of intraocular pressure lowering medication within the past 3 months or any history of ocular surgery for glaucoma
* Evidence of potential angle closure by gonioscopy
* Abnormal optic disc or visual field consistent with glaucoma
* Use of topical ocular medications during the study and any evidence of systemic disease that might interfere with the conduct of the study.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 54 (Actual)
Dates: Start 2007-10; Primary Completion 2008-08 (Actual); Study Completion 2008-10 (Actual)

PRIMARY OUTCOMES:
The reduction of IOP as calculated on the basis of the arithmetic mean of up to six measurements of IOP, comparing baseline to visit 6 | 28 days of therapy

SECONDARY OUTCOMES:
Percentage change and responder rates - e.g., > 20% reduction in lOP values from baseline to Day 21, Day 14 and Day 7 | 7, 14, 21 days of therapy

CONTACTS AND LOCATIONS:
Overall Officials: Barrett Katz, MD, Study Chair — CEO, CMO, Danube Pharmaceuticals, Inc.
Locations (1):
- Omnicare Clinical Research Center, Chippenham, Wiltshire, United Kingdom